CLINICAL TRIAL: NCT05321953
Title: The Impact of Aerobic Interval and Inspiratory Muscle Training On Patient Reported Constipation Outcome Scores In Individuals With Chronic Constipation Who Plateau or Are Non- Responders to Biofeedback Therapy: A Call to Treat Beyond The Pelvic Floor
Brief Title: The Impact of Aerobic Interval and Inspiratory Muscle Training On Patient Reported Outcome Scores In Individuals With Chronic Constipation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: University of Miami (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Lawrence Cahalin, Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210958
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-06

CONDITIONS: Constipation; Constipation by Outlet Obstruction; Constipation-predominant Irritable Bowel Syndrome; Constipation - Functional
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Physical Therapy With No Study Intervention (Active Comparator): Participants will receive 6 weeks of standard physical therapy and have reported satisfaction and respond with a numerical value of ≤3 on a chronic constipation numeric scale. Participants will receive no additional study interventions.
  Interventions: Other: Standard Physical Therapy Care
- Standard of Care Physical Therapy With Study Intervention (Experimental): Participants who receive 6 weeks of standard physical therapy and have reported non satisfaction and respond with a numerical value of >3 on a chronic constipation numeric scale and have been cleared of pelvic floor muscle dyssynergia. Participants will receive an additional 8 weeks of study intervention.
  Interventions: Other: Standard Physical Therapy Care; Other: Aerobic and Inspiratory Muscle Training

INTERVENTIONS:
Other: Standard Physical Therapy Care — Standard physical therapy care. Six to eight, one hour sessions over the course of 4-6 weeks. For individuals with chronic constipation that includes biofeedback therapy, breathing techniques on the toilet, manual therapy to the abdominal wall, and education on toileting posture and favorable lifestyle habits for gut health.
Other: Aerobic and Inspiratory Muscle Training — The exercise-based 3 times per week for 8 weeks intervention will consist of aerobic interval training and inspiratory muscle training (IMT) for a total duration of 30 minutes. Aerobic-based intervals will be performed at a moderate intensity. Aerobic modes of exercise will include upper extremity ergometer, treadmill, bike, or elliptical.
  Arms: Standard of Care Physical Therapy With Study Intervention

SUMMARY:
The primary aim of this study will be to determine if the addition of aerobic interval and inspiratory muscle training (IMT) targeted at improving cardiopulmonary-based measures will further improve patient satisfaction scores in individuals with chronic constipation (CC) who report plateau or limited improvements in CC after demonstrating a corrected defecation pattern using anorectal biofeedback training.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Complaint of chronic constipation and associated symptoms
* Confirmed pelvic floor muscle dyssynergia
* Willing and able to sign informed consent
* Ability to comply with study guidelines.
* Potential subjects must report two or more of the following: straining during more than 25% of defecations, lumpy or hard stools more than 25% of defecations, sensations of incomplete bowel evacuation more than 25% of defecations, manual maneuvers to facilitate more than 25% of defecations, sensation of anorectal obstruction/blockage more than 25% of defecations, and fewer than 3 small bowel movements per week.

Exclusion Criteria:

* Rectal prolapse greater than grade 2
* Pregnancy
* Cognitive impairments
* History or present cardiac condition that would exclude them from moderate intensity exercise
* Presence of an orthopedic condition with significant severity that the exercise protocol may exacerbate
* Currently receiving additional physical therapy treatment for conditions associated with pelvic floor muscle dysfunction
* Recent surgery within the past 3 months without clearance from a medical doctor
* Medication usage that would interfere with their ability to exercise safely
* Individuals recovering from a confirmed eating disorder or recent unexplained weight loss >10lbs within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Change In Patient Assessment of Constipation Symptoms (PAC-SYM) | Baseline, 6 weeks, 14 weeks, 26 weeks
  The PAC-SYM questionnaire is a 12 item questionnaire that consists of three subscales: abdominal, rectal, and stool. Each item is scored 0-4 (0: Absent, 1: Mild, 2: Moderate, 3: Severe, 4: Very Severe). A total raw score can range from 0-48. The final score is the average of the summed score divided by the number of items, ranging from 0: Absent, 1: Mild, 2: Moderate, 3: Severe, 4: Very Severe.

SECONDARY OUTCOMES:
Change In Distance by the Incremental Shuttle Walk Test (ISWT) | Week 6, week 14
  The Incremental Shuttle Walk Test (ISWT) is an incremental externally paced walking test and is generally used as an index of cardiorespiratory fitness. The primary outcome is the distance covered calculated from the completed number of shuttles. The ISWT distance can be used to track changes in exercise capacity over time.
Change In estimated oxygen consumption (eVO2) by the Incremental Shuttle Walk Test (ISWT) | Week 6, week 14
  The Incremental Shuttle Walk Test (ISWT) is an incremental externally paced walking test and is generally used as an index of cardiorespiratory fitness. Peak estimated oxygen consumption (eVO2) can be estimated with greater accuracy than other field tests using a linear prediction equation incorporating ISWT distance.
Change In Heart Rate Recovery (HRR) | Week 6, week 14
  Heart rate recovery (HRR) will be measured as the difference of the peak heart rate at the end of the first exercise session and one minute post exercise. This will be recorded through the Polar Heart Rate chest monitor.
Change In Maximal Inspiratory Pressure (PImax) | Week 6, week 14
  PImax will be measured via the test of incremental respiratory endurance (TIRE) using the Pro2fit device and application.
Change In Rand Short Form Health Survey Questionnaire (SF-36) scores | Week 6, week 14
  The SF-36 is a widely recognized outcome measure used to measure health status in a variety of populations. The measure consists of eight domains and each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Lower scores measure more disability and higher scores measure less disability. Scores represent the percentage of the total possible score achieved. Items in the same domain are averaged together to create 8 scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cahalin, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No